CLINICAL TRIAL: NCT01434017
Title: Comparison of Three Different Prophylactic Treatments of PONV in Children
Brief Title: Comparison of Three Different Prophylactic Treatments of Postoperative Nausea and Vomiting (PONV) in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Eric Albrecht, MD, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CHUV-51-08
Record Dates: First submitted 2011-09-13; First posted 2011-09-14 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-02

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: PONV; Dexamethasone; Droperidol; Ondansetron; Tonsillectomy
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Dexamethasone; Droperidol; Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dexamethasone (Active Comparator): Patients will receive dexamethasone 250 mcg/kg just after induction of anesthesia.
  Interventions: Drug: Dexamethasone
- Dexamethasone and Droperidol (Active Comparator): Patients will receive dexamethasone 250 mcg/kg + droperidol 10 mcg/kg just after induction of anesthesia.
  Interventions: Drug: Dexamethasone and droperidol
- Dexamethasone and Ondansetron (Active Comparator): Patients will receive dexamethasone 250 mcg/kg + ondansetron 150 mcg/kg just after induction of anesthesia.
  Interventions: Drug: Dexamethasone and Ondansetron

INTERVENTIONS:
Drug: Dexamethasone — Patients will receive dexamethasone 250 mcg/kg just after induction of anesthesia.
  Arms: Dexamethasone
Drug: Dexamethasone and droperidol — Patients will receive dexamethasone 250 mcg/kg + droperidol 10 mcg/kg just after induction of anesthesia.
  Arms: Dexamethasone and Droperidol
Drug: Dexamethasone and Ondansetron — Patients will receive dexamethasone 250 mcg/kg + ondansetron 150 mcg/kg just after induction of anesthesia.
  Arms: Dexamethasone and Ondansetron

SUMMARY:
Incidence of postoperative nausea and vomiting (PONV) in children after tonsillectomy with or without adenoidectomy may be as high as 75%.

Several medications may prevent and treat PONV, such as steroids, antidopaminergic drugs and serotonin (5-HT3) antagonists. The objective of this study is to compare three prophylactic antiemetic treatments:

* dexamethasone alone (250 mcg/kg)
* dexamethasone (250 mcg/kg) + droperidol (10 mcg/kg)
* dexamethasone (250 mcg/kg) + ondansetron (150 mcg/kg).

DETAILED DESCRIPTION:
Tonsillectomy with or without adenoidectomy may be associated with severe postoperative nausea and vomiting (PONV). Causes are principally trigeminal nerve stimulation and presence of blood in the stomach. Consequences are disagreement, unsatisfactory, delayed discharge, and overnight admission in day-cases. More barely, patients may also have suture and esophagus rupture, aspiration of gastric contents, dehydration and electrolyte disturbances.

Several medications may prevent and treat PONV, such as steroids, antidopaminergic drugs and serotonin (5-HT3) antagonists. The objective of this study is to compare three prophylactic antiemetic treatments:

* dexamethasone alone (250 mcg/kg)
* dexamethasone (250 mcg/kg) + droperidol (10 mcg/kg)
* dexamethasone (250 mcg/kg) + ondansetron (150 mcg/kg).

The hypothesis is that the combination of dexamethasone and droperidol is as effective as the combination of dexamethasone and ondansetron, both of them being more effective than dexamethasone alone. Moreover, droperidol is cheaper than ondansetron and may be recommended as a first-line treatment.

ELIGIBILITY:
Inclusion Criteria:

* children aged 2-10 y.
* children ASA 1-2
* weight > 15 kg
* tonsillectomy with or without adenoidectomy

Exclusion Criteria:

* intravenous induction
* contraindication to steroids
* contraindication to antidopaminergic drugs
* contraindication to serotoninergic antagonists
* administration of steroids, antidopaminergic drugs, or serotoninergic antagonists in the 24 hours before the surgery
* refusal of parents
* no-french speaking parents

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2008-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Incidence of PONV after tonsillectomy with or without adenoidectomy | 48 hours

SECONDARY OUTCOMES:
Incidence of side effects (extrapyramidal syndrome, hemorrhage, somnolence, headaches) | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Eric Albrecht, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (1):
- Centre Hospitalier Universitaire Vaudois and University of Lausanne, Lausanne, Canton of Vaud, Switzerland